CLINICAL TRIAL: NCT04799392
Title: NOWDx Test for the Detection of Antibodies to COVID-19 in Lay Persons
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA will not authorize COVID-19 Ab tests for use over-the-counter.
Sponsor: NOWDiagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NOWDx COVID-19 Antibody OTC
Record Dates: First submitted 2021-03-14; First posted 2021-03-16 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Persons tested with investigational device following PCR test (Experimental): Persons tested with investigational device who previously tested positive or negative for COVID-19 with an emergency use authorized or FDA cleared COVID-19 test
  Interventions: Device: NOWDx COVID-19 Test
- Persons tested with investigational device following vaccination (Experimental): Persons tested with investigational device who previously were vaccinated for COVID-19 with an emergency use authorized or FDA cleared COVID-19 vaccine
  Interventions: Device: NOWDx COVID-19 Test

INTERVENTIONS:
Device: NOWDx COVID-19 Test — The investigational device is the NOWDx COVID-19 Test.

SUMMARY:
This study is designed to compare the performance of the NOWDx COVID-19 Test to an emergency use authorized PCR test result. The intent is to show the rapid test device is comparable to a currently marketed device. The NOWDx COVID-19 Test is an in vitro lateral flow immunoassay intended for qualitative detection of total antibodies to SARS-CoV-2 in human fingerstick whole blood at the Point of Care (POC); i.e. in patient care settings operating under a CLIA Certificate of Waiver, Certificate of Compliance, or Certificate of Accreditation; and at home.

DETAILED DESCRIPTION:
This study is designed to compare the performance of the NOWDx COVID-19 Test to an emergency use authorized PCR test result. The intent is to show the rapid test device is comparable to a currently marketed device. The NOWDx COVID-19 Test is an in vitro lateral flow immunoassay intended for qualitative detection of total antibodies to SARS-CoV-2 in human fingerstick whole blood at the Point of Care (POC); i.e. in patient care settings operating under a CLIA Certificate of Waiver, Certificate of Compliance, or Certificate of Accreditation; and at home.

The NOWDx COVID-19 Test is intended for use as an aid in identifying individuals with an adaptive immune response to SARS-CoV-2, indicating recent or prior infection. At this time, it is unknown for how long antibodies persist following infection and if the presence of antibodies confers protective immunity. Testing of human fingerstick whole blood is intended to be conducted in a home-like setting of a facility authorized to perform CLIA waived tests.

ELIGIBILITY:
Inclusion Criteria:

Innate Infection Cohort>

* PCR positives: persons who were symptomatic for COVID-19 and have tested positive for COVID-19 with an EUA or FDA cleared PCR test; 7+ days post positive PCR test
* PCR negatives: persons who have never had COVID-19 and who have tested negative for COVID-19 with an EUA or FDA cleared PCR test; within 0-6 days post negative PCR test
* persons 2+ years old

Vaccination Cohort>

* persons 7- 60 days post second dose of EUA COVID-19 vaccine
* persons 18+ years old

Exclusion criteria:

Innate Infection Cohort>

* PCR positives: persons with a COVID-19 positive test result >45 days old
* PCR negatives: persons with any prior COVID-19 positive result
* persons who have received COVID-19 vaccine
* persons <2 years old

Vaccination Cohort>

* persons symptomatic or previously infected with COVID-19 prior to vaccination
* persons <18 years old

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Percentage of clinical agreement between NOWDx COVID-19 Test and emergency use authorized or FDA cleared comparator | through study completion; an average of 2 months
  Calculate positive percent agreement (PPA) and negative percent agreement (NPA) between NOWDx COVID-19 Test and emergency use authorized or FDA cleared COVID-19 PCR test.
Positivity rate of NOWDx COVID-19 Tests in vaccinated persons | through study completion; an average of 2 months
  Calculate positivity rate of NOWDx COVID-19 Tests in persons post emergency use authorized or FDA cleared COVID-19 vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Cobb, Principal Investigator — NOW Diagnostics, Inc.
Locations (5):
- United States (5):
  - Medical Arts Pharmacy, Fayetteville, Arkansas
  - Goodrich Pharmacy, Anoka, Minnesota
  - Alps Specialty Pharmacy, Nixa, Missouri
  - Alps Pharmacy, Springfield, Missouri
  - Bremo Pharmacy, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No